CLINICAL TRIAL: NCT05555680
Title: Effect of Hyperandrogenism on IVF Success Rates in PCOS Patients
Brief Title: Effect of Hyperandrogenism on IVF Outcomes in PCOS Patients
Acronym: HIP
Status: Terminated | Type: Observational
Why Stopped: Low recruitment rate
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: CCER 21-22 - 31
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
Keywords: Hyperandrogenism; Fertility issues
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS patients with clinical or biochemical hyperandrogenism: Clinical hyperandrogenism consists of patients with one of the following conditions: Acne, Hirsutism (using modified Ferriman-Gallwey (FG) score) or Androgenic alopecia Biochemical hyperandrogenism consists of elevated serum level of at least one of the following hormones: Total testosterone, free testosterone, DHEAS, androstenedione using the cut-offs adopted by the laboratory.
  Interventions: Other: Ferriman-Gallwey Score
- PCOS patients with no clinical or biochemical hyperandrogenism: In this cohort, women have not be affected by either clinical of biochemical hyperandrogenism. The PCOS diagnosis will be based on oligo-anovulation and on polycystic ovaries during an ultrasound
  Interventions: Other: Ferriman-Gallwey Score

INTERVENTIONS:
Other: Ferriman-Gallwey Score — The Ferriman-Gallwey score is used to evaluate hirsutism. The examiner scores the subjects on a scale of 0-4 for terminal hair growth on eleven different body areas according to the Ferriman-Gallwey scoring system. A Ferriman-Gallwey score of 8 or more was considered diagnostic of hirsutism

SUMMARY:
Ovulatory dysfunction affects 18 to 25% of infertile women, the most common identifiable condition is polycystic ovarian syndrome (PCOS). The most frequent symptoms of PCOS are oligo-anovulation, hyperandrogenism and polycystic ovary appearance.

Hyperandrogenism is the main contributor that affects oocyte and embryo quality and decreases the success rates in PCOS patients undergoing IVF treatments.

The aim of this study is to determine the effect of hyperandrogenism as an independent factor on IVF success rates and oocyte/embryo quality in PCOS patients undergoing IVF.

DETAILED DESCRIPTION:
Despite that PCOS patients obtain a higher yield of oocytes retrieved in IVF treatments, they often have lower fertilization, cleavage and implantation rates and a higher rate of miscarriage, which can be attributed to a poor quality of retrieved oocytes and the resulting embryos. Multiple studies compared IVF outcomes in PCOS patients to control groups and found that PCOS might negatively affect oocyte maturation rate, fertilization rate in conventional IVF and miscarriage rate. Hence, it seems that PCOS might be associated with poor outcomes in IVF cycles when compared to non-PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* Women between ages of 18 - 39 inclusively
* ≥15 oocytes collected on the day of oocyte retrieval and/or anti-mullerian hormone (AMH) ≥ 4.0 ng/ml in the participant's medical chart in the last 24 months

Exclusion Criteria:

* Male factor necessitating testicular sperm aspiration (TESA), testicular sperm extraction (TESE) or micro-TESE
* Fertility preservation
* Recurrent pregnancy losses (RPL) (defined as 2 or more failed clinical pregnancies as documented by ultrasonography or histopathologic examination,or 3 or more failed pregnancies before 14 weeks of gestation)
* Oocyte donation
* Medical diagnosis of non classic congenital adrenal hyperplasia diagnosed based on 17 hydroxyprogesterone level

Ages: 18 Years to 39 Years | Sex: Female
Age Groups: Adult
Study Population: PCOS patients undergoing the first embryo transfer following the first IVF treatment during the study period (or up to two embryo transfers)
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of hyperandrogenism on frozen embryo transfer | 10 days after frozen embryo transfer
  Determine the effect of PCOS subjects affected by hyperandrogenism (HA) on clinical pregnancy rate following a frozen embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Benoit, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No